CLINICAL TRIAL: NCT03641313
Title: A Phase 2 Single-Arm Study of M6620 in Combination With Irinotecan in Patients With Progressive TP53 Mutant Gastric and Gastro-Esophageal Junction Cancer
Brief Title: Berzosertib and Irinotecan in Treating Patients With Progressive, Metastatic, or Unresectable TP53 Mutant Gastric or Gastroesophageal Junction Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01739; NCI-2018-01739 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC LOI#18012; 10211 (Other: Yale University Cancer Center LAO); 10211 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Unresectable Gastric Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — berzosertib; Endoscopic Mucosal Resection; Endoscopy; Biopsy; Irinotecan; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (irinotecan and M6620) (Experimental): Patients receive irinotecan IV over 90 minutes and berzosertib IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo endoscopic or CT assisted biopsy and MRI on study.
  Interventions: Drug: Berzosertib; Procedure: Computed Tomography Assisted Biopsy; Procedure: Endoscopic Biopsy; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Procedure: Computed Tomography Assisted Biopsy — Undergo CT assisted biopsy
  Other Names: Computed Tomography Biopsy; Computed Tomography-Guided Needle Biopsy; CT Assisted Biopsy; CT Guided Biopsy
Procedure: Endoscopic Biopsy — Undergo endoscopic biopsy
  Other Names: Endoscopy and Biopsy
Drug: Irinotecan — Given IV
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial studies the how well berzosertib and irinotecan work in treating patients with gastric or gastroesophageal junction cancer that is growing, spreading or getting worse (progressive), has spread to other places in the body (metastatic), or cannot be removed by surgery (unresectable). Berzosertib may stop the growth of tumor cells by blocking some of the enzymes needed for growth. Chemotherapy drugs, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving berzosertib and irinotecan may work better than irinotecan alone in treating patients with gastric and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine objective response rate (ORR) superiority (target 25%) in TP53 mutant patients with progressive metastatic or unresectable gastric/gastroesophageal junction (GEJ) cancer who receive berzosertib (M6620) and irinotecan compared to ORR (5%) in historical control patients treated with single agent irinotecan alone.

SECONDARY OBJECTIVES:

I. Determine duration of response (DOR), time to progression (TTP), progression-free survival (PFS), and overall survival (OS) superiority in TP53 mutant gastric/GEJ cancer patients who receive M6620 and irinotecan compared to these measures in historical control patients treated with irinotecan alone.

II. Perform the following correlative studies in 9 patients: gamma-H2AX, KAP1 phosphorylated (p)-Ser 824 and p-ATR analysis from biopsies collected at 24 hours (+/- 1 hour) post-irinotecan infusion on cycle 1 day 2 (C1D2) and at 24 hours (+/- 1 hour) post-M6620 on cycle 2 day 2 (C2D2).

EXPLORATORY OBJECTIVES:

I. Determine ORR, DOR, TTP, PFS, and OS in patients with other concomitant damage response defects (DDRD), such as mutations in BRCA1, BRCA2, MRE11, RAD50, RAD51, RAD52, RAD54L, NBN, ATM, H2AX, PALB2, RPA, BRIP1, BARD1, ATR, ATRX, CHK1, CHK2, MDM2, MDM4, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCL, treated with the experimental combination.

II. Determine whether patients with first line platinum sensitivity (PFS > 3 months) demonstrate improved ORR, DOR, TTP, PFS, and OS compared to patients who were platinum insensitive (PFS < 3 months).

OUTLINE:

Patients receive irinotecan intravenously (IV) over 90 minutes and berzosertib IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo endoscopic or computed tomography (CT) assisted biopsy and magnetic resonance imaging (MRI) on study.

After completion of study treatment, patients are followed up for 30 days and then every 2 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed progressive metastatic or unresectable gastric or GEJ adenocarcinoma.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Patients must have progressed after or been intolerant of at least two lines of systemic therapy. Patients with HER2 positive gastric and GEJ adenocarcinoma must have progressed on trastuzumab plus chemotherapy in the first line setting. Patients with microsatellite unstable (MSI-H) tumors must have received prior immunotherapy with pembrolizumab.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M6620 in combination with irinotecan in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Both men and women of all races and ethnic groups are eligible for this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 60%).
* Leukocytes >= 3,000/mcL.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 100,000/mcL.
* Hemoglobin >= 9 g/dL.
* Total bilirubin within normal institutional limits.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN); if liver involvement =< 5 x ULN.
* Creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Patients must have a TP53 mutation (only those known hot-spot mutations that fall within exon 2 or exons 4-11 will be accepted) determined from available archived tumor tissue that has been subjected to next generation sequencing (NGS) through FoundationOne/FoundationOneCDx or a similar assay performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. Investigators from other sites, who have potential patients who meet study eligibility, will send copies of NGS reports from these patients via Medidata Rave case reports to the responsible study coordinator. Our research team will review each report to ensure each patient possesses the mutations of interest. Similar review will happen for each patient we enroll on the study at our institution. Case reports from all screened patients will be centrally available on the Rave study database.
* Nine patients must be willing to undergo endoscopic or CT guided tumor biopsies for mandatory correlative studies. If the biopsy is deemed not safe by the treating physician, the patient may still enroll given that the other eligibility criteria are met.
* The effects of M6620 on the developing human fetus are unknown. For this reason and because deoxyribonucleic acid (DNA)-damage response (DDR) inhibitors, as well as irinotecan, are known to be teratogenic, women of child-bearing potential and men able to father children who have female partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after trial participant's final dose of M6620 or irinotecan (whichever agent is completed last). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with early stage untreated or resectable gastric adenocarcinoma.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients who have previously received irinotecan.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1, except alopecia) that was administered more than four weeks prior to starting study therapy.
* Patients who are receiving any other investigational agents.
* Patients with untreated or symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 or irinotecan.
* M6620 is primarily metabolized by CYP3A4, and irinotecan and its active metabolite, SN-38, are metabolized by CYP3A4 and UGT1A1, respectively; therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) or inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) should be avoided. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because M6620 as a DNA-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620, breastfeeding should be discontinued if the mother is treated with M6620. These potential risks also apply to irinotecan.
* Human immunodeficiency virus (HIV)-positive patients are excluded unless they have an undetectable viral load and are able to use anti-viral agents that do not interact with CYP3A4 (or regimens with agents that are not major inhibitors of cytochrome P450 enzymes).
* History of other malignancy within 36 months prior to enrollment. Patients with local cancers of any type, provided no recurrence over this timeframe, are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-01-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Berlin, Principal Investigator — Yale University Cancer Center LAO
Locations (31):
- United States (31):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Wheless MC, Stockton S, Soares HP, Dayyani F, Saeed A, Kim E, Jin N, Yacoub G, Florou V, Ayers GD, Guerrouahen BS, Contreras A, Li L, Ferry-Galow KV, Gore S, Das S, Berlin J. NCI 10211: a phase II, single-arm study of berzosertib in combination with irinotecan in patients with advanced TP53 mutant gastroesophageal cancer. Oncologist. 2025 Dec 1;30(12):oyaf400. doi: 10.1093/oncolo/oyaf400. PMID 41335461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from participating academic medical centers within the Experimental Therapeutics Clinical Trials Network (ETCTN) between 30-Jun-2020 and 01-Dec-2022.
Period: Overall Study
Arm/Group | Treatment (Irinotecan and M6620)
Started (Study consented 19 patients but 2 were screen fails and did not start treatment.) | 17 (Participants started treatment)
Completed | 12
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Declining health | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 76]
Number of participants included in primary endpoint of objective response rate [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Response Criteria
Description: Number of patients that achieved either a partial response or complete response as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 response criteria. Per RECIST v.1.1 assessed by CT or MRI: complete response (CR) is disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Overall response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Duration of Responses (DOR)
Description: As 0 participants achieved a response (either complete response or partial response), data for this outcome measure can not be calculated.
Time Frame: From when patients achieve their best response (complete response [CR] or partial response [PR]) to when they progress or die for any reason, assessed up to 1 year
Population: As 0 participants achieved a response (either complete response or partial response), data for this outcome measure can not be calculated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
months | NA [NA to NA] — As 0 participants achieved a response (either complete response or partial response), data for this outcome measure can not be calculated.

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression was calculated for all participants. Progression was defined as: 1) using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions; and 2) clinical progression as defined by participant's treating physician. This measure was estimated using the method of Kaplan and Meier and presented with 95% confidence intervals.
Time Frame: From start of treatment to time of progression or death from progression, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
months | 3.5 [1.8 to 4.8]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was calculated for all participants. Progression was defined as: 1) using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions; and 2) clinical progression as defined by participant's treating physician. This measure was estimated using the method of Kaplan and Meier and presented with 95% confidence intervals.
Time Frame: From enrollment to disease progression or death for any reason, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
months | 4.01 [2.07 to NA] — NA means that he upper 95% confidence interval was not reached

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was calculated for all participants. Will be estimated using the method of Kaplan and Meier and presented with 95% confidence intervals.
Time Frame: From study enrollment to death for any reason, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Irinotecan and M6620)
Number analyzed (Participants) | 17
months | 6.21 [4.83 to 8.61]

6. Other Pre Specified Outcome: ORR in Sub-cohorts Based on First-line Platinum Sensitivity
Description: Number of participants that had a partial response or complete response to treatment per RECIST v1.1 categorized by platinum sensitivity. Platinum sensitivity was defined as receiving a prior platinum-based therapy for more than 3 months. Per RECIST v.1.1 assessed by CT or MRI: complete response (CR) is disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Overall response (OR) = CR + PR.
Time Frame: Up to 1 year
Population: Three of the 17 patients did not have available prior treatment data to determine if they were platinum sensitive or not sensitive.
Measure: Count of Participants; unit: Participants
Groups:
- Platinum Sensitive: Patients that were on a prior platinum containing regimen for longer than 3 months.
- Platinum Not Sensitive: Patients that has progressive disease within 3 months on a prior platinum-based treatment regimen
Arm/Group | Platinum Sensitive | Platinum Not Sensitive
Number analyzed (Participants) | 10 | 4
Participants | 0 | 0

7. Other Pre Specified Outcome: DOR in Sub-cohorts Based on First-line Platinum Sensitivity
Description: as for outcome 2
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Platinum Sensitive | Platinum Not Sensitive
Number analyzed (Participants) | 10 | 4
months | NA [NA to NA] — As 0 participants achieved a response (either complete response or partial response), data for this outcome measure can not be calculated. | NA [NA to NA] — As 0 participants achieved a response (either complete response or partial response), data for this outcome measure can not be calculated.

8. Other Pre Specified Outcome: TTP in Sub-cohorts Based on First-line Platinum Sensitivity
Description: Time to progression was calculated for sub cohorts of participants based on sensitivity to prior platinum-based treatment. Progression was defined as: 1) using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions; and 2) clinical progression as defined by participant's treating physician. This measure was estimated using the method of Kaplan and Meier and presented with 95% confidence intervals.
Time Frame: Up to 1 year
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Platinum Not Sensitive: Patients that had progressive disease within 3 months on a prior platinum-based treatment regimen
Arm/Group | Platinum Sensitive | Platinum Not Sensitive
Number analyzed (Participants) | 10 | 4
months | 4.3 [1.7 to NA] — NA means that he upper 95% confidence interval was not reached | 1.9 [1.8 to NA] — NA means that he upper 95% confidence interval was not reached

9. Other Pre Specified Outcome: PFS in Sub-cohorts Based on First-line Platinum Sensitivity
Description: Progression-free survival was calculated for sub cohorts of participants based on sensitivity to prior platinum-based treatment. Progression was defined as: 1) using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions; and 2) clinical progression as defined by participant's treating physician. This measure was estimated using the method of Kaplan and Meier and presented with 95% confidence intervals.
Time Frame: Up to 1 year
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Platinum Sensitive | Platinum Not Sensitive
Number analyzed (Participants) | 10 | 4
months | 4.0 [1.7 to 4.8] | 1.9 [1.8 to NA] — NA means that he upper 95% confidence interval was not reached

10. Other Pre Specified Outcome: OS in Sub-cohorts Based on First-line Platinum Sensitivity
Description: Overall survival was calculated for sub cohorts of participants based on sensitivity to prior platinum-based treatment
Time Frame: Up to 1 year
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Platinum Sensitive | Platinum Not Sensitive
Number analyzed (Participants) | 10 | 4
months | 6.2 [3.7 to 7.2] | 4.4 [2.1 to NA] — NA means that he upper 95% confidence interval was not reached

11. Other Pre Specified Outcome: Presence of Other Deoxyribonucleic Acid (DNA) Damage Response Defects (DDRD)
Description: Mutations present will be summarized as frequency counts and percent of study group.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- ATRX Mutation: Count of participants with an ATRX mutation
- MDM2 Mutation: Count of participants with an MDM2 mutation
Arm/Group | ATRX Mutation | MDM2 Mutation
Number analyzed (Participants) | 17 | 17
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events that emerge (or worsen) after the first dose of study drug and within 30 days after the last dose.
Arm/Group | Treatment (Irinotecan and M6620)
All-Cause Mortality (participants affected / at risk) | 17/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Irinotecan and M6620) (N=17)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Irinotecan and M6620) (N=17)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphatase increased (Investigations) | 5 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (20)
Anemia (Blood and lymphatic system disorders) | 9 (53)
Anorexia (Metabolism and nutrition disorders) | 6 (14)
Anxiety (Psychiatric disorders) | 2 (9)
Ascites (Gastrointestinal disorders) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (4)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bubbling saliva (Gastrointestinal disorders) | 1 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Cholinergic reaction (Immune system disorders) | 1 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Creatinine increased (Investigations) | 2 (11)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (50)
Dizziness (Nervous system disorders) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ear fullness bilateral (Ear and labyrinth disorders) | 1 (8)
Edema limbs (General disorders) | 3 (10)
Elevated eGFR (Renal and urinary disorders) | 1 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 8 (26)
Fever (General disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Gastroparesis (Gastrointestinal disorders) | 1 (6)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (13)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (24)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 6 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (10)
Hypotension (Vascular disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Inflamed seborrheic keratosis on upper chest (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (8)
Lymphocyte count decreased (Investigations) | 7 (39)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muffled hearing (Ear and labyrinth disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (5)
Nausea (Musculoskeletal and connective tissue disorders) | 12 (42)
Neutrophil count decreased (Investigations) | 6 (6)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (15)
Platelet count decreased (Investigations) | 2 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Pyelonephritis (Infections and infestations) | 1 (1)
Red bump on abdomen (Skin and subcutaneous tissue disorders) | 1 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sepsis (Infections and infestations) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (8)
Urinary frequency (Renal and urinary disorders) | 1 (4)
Urinary retention (Renal and urinary disorders) | 1 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (25)
Weight loss (Infections and infestations) | 2 (7)
White blood cell decreased (Infections and infestations) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03641313/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03641313/ICF_001.pdf